CLINICAL TRIAL: NCT06748794
Title: Effects of Intrathecal Midazolam (1mg) With Hyperbaric Bupivacaine 0.5% (15mg) for Spinal Anesthesia for Caesarean Section
Brief Title: Effects of Intrathecal Midazolam (1mg) With Hyperbaric Bupivacaine 0.5% (15mg) for Spinal Anesthesia for C-section
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/049
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Chromosomes, Human, 1-3

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: group 1 — A comparative analysis was conducted to assess sensory and motor block characteristics, postoperative analgesia duration, maternal hemodynamic stability, and neonatal outcomes. Results demonstrated that intrathecal midazolam significantly prolonged postoperative analgesia and reduced analgesic requirements while maintaining hemodynamic stability and maternal-neonatal safety. This combination provides a potential enhancement to spinal anesthesia techniques, improving maternal comfort and overall perioperative outcomes in obstetric patients.

SUMMARY:
This study evaluates the effects of intrathecal midazolam (1 mg) combined with hyperbaric bupivacaine 0.5% (15 mg) for spinal anesthesia in cesarean section patients.

DETAILED DESCRIPTION:
The addition of midazolam, a benzodiazepine with analgesic and anxiolytic properties to bupivacaine is hypothesized to enhance the quality of anesthesia and postoperative pain relief without significant side effects. A comparative analysis was conducted to assess sensory and motor block characteristics, postoperative analgesia duration, maternal hemodynamic stability, and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female patients presented for elective cesarean section.
* All ASA I & II patients .
* Age between 18 to 35 years.

Exclusion Criteria:

* Contraindication to spinal anesthesia.
* Patient not willing or previous bad experience with it.
* All ASA III & IV class was excluded from the study.
* Patients with documented bleeding disorders i.e. low platelet count, deranged PT/APTT/INR, DIC etc.
* Hypertensive patients
* Patients with Diabetes mellitus.
* Obese patients BMI >30.
* PIH (pre- eclampsia and eclapmsia)"

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Caesarean Section
Study Population: to check the Effects of Intrathecal Midazolam (1mg) With Hyperbaric Bupivacaine 0.5% (15mg) for Spinal Anesthesia for Caesarean Section
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 12 Months
  Time from intrathecal drug administration to the first request for additional analgesia by the patient.
Quality of sensory and motor block | 12 Months
  Onset, level, and duration of sensory block, Onset and duration of motor block, Maximum sensory block level achieved.
Hemodynamic stability | 12 months
  Incidence and severity of hypotension, bradycardia, or other hemodynamic changes during the perioperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- Nowshera, Nowshera, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No